CLINICAL TRIAL: NCT06732258
Title: Exploratory Clinical Study of Low-dose Radiotherapy Combined with Concurrent Chemotherapy, Toripalimab and Tifcemalimab in First-line Treatment of Extensive-Stage Small Cell Lung Cancer
Brief Title: Low-dose Radiotherapy Combined with Concurrent Chemotherapy, Toripalimab and Tifcemalimab in the Treatment of ES-SCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONTEST
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: ES-SCLC; Toripalimab; Tifcemalimab; LDRT
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Radiotherapy; toripalimab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose radiotherapy concurrent Chemotherapy combined with Toripalimab and Tifcemalimab (Experimental)
  Interventions: Radiation: Low-dose radiotherapy; Drug: Tifcemalimab injection; Drug: Toripalimab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Radiation: Low-dose radiotherapy — The LDRT deals with primary tumour in a 15 Gy of 5 fractions over five days, starting from Day 1 in the first cycle.
Drug: Tifcemalimab injection — 100 mg or 200 mg q3w until disease progression or intolerable toxicity;
Drug: Toripalimab — 240 mg q3w until disease progression or intolerable toxicity;
Drug: Cisplatin — 75 mg/m2 q3w for 4-6 cycles;
Drug: Carboplatin — AUC = 5, q3w for 4-6 cycles;
Drug: Etoposide — 100 mg/m2, d1, d2, d3, q3w for 4-6 cycles;

SUMMARY:
To evaluate the tolerability and safety of Low-dose radiotherapy combined with concurrent Chemotherapy, Toripalimab and Tifcemalimab in first-line treatment of Extensive-Stage Small Cell Lung Cancer, and to determine the RP2D.

DETAILED DESCRIPTION:
This is a single-center, single-arm, exploratory clinical study to evaluate the safety and tolerability of low-dose radiotherapy (LDRT) concurrent chemotherapy combined with toripalimab and Tifcemalimab (JS004) in the first-line treatment of extensive-stage small cell lung cancer (ES-SCLC). Approximately 6-12 subjects were planned to be enrolled in this clinical study. The study will adopt a "3 + 3" dose escalation design, and the observation period for dose-limiting toxicities (DLTs) is 21 days after the first dose administration. Patients who meet the inclusion criteria will receive toripalimab 240 mg q3w, tifcemalimab 100 mg or 200 mg q3w until disease progression or intolerable toxicity; cisplatin for injection 75 mg/m2 or carboplatin AUC = 5, q3w, etoposide 100 mg/m2, d1, d2, d3, q3w for 4-6 cycles; low-dose radiotherapy with a total dose of 15 Gy, radiotherapy will be started on Cycle 1 Day 1 in 5 divided doses (15 Gy/5F).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female;
* Histologically or cytologically confirmed extensive stage small cell lung cancer;
* Previously untreated extensive stage small cell lung cancer;
* ECOG PS 0-1;
* Measurable lesions according to RECIST 1.1, and measurable lesions can only be included in previously irradiated lesions if the lesion shows definite disease progression after radiotherapy;
* Expected survival ≥ 3 months;
* Normal function of major organs, that is, meet the following criteria: neutrophils ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, hemoglobin ≥ 90 g/L; serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min; serum total bilirubin ≤ 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; ALT and AST ≤ 5 × ULN in patients with liver metastases; international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN unless the subject is receiving anticoagulant therapy, activated partial thrombin time (aPTT) ≤ 1.5 × ULN unless the subject is receiving anticoagulant therapy;
* Female subjects of childbearing potential, as well as male subjects with partners of childbearing potential, need to use a medically recognized contraceptive (such as an intrauterine device, contraceptive, or condom containing spermicide) during study treatment and for at least 4 months after the last use of study drug;
* Voluntary participation in this study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

* Mixed SCLC and non-small cell lung cancer (NSCLC);
* Symptomatic, untreated or progressive central nervous system (CNS) metastases;
* Received any systemic anti-tumor therapy for ES-SCLC;
* Previously received any immune checkpoint inhibitors, including but not limited to CTLA-4 inhibitors, PD-1/PD-L1 inhibitors, BTLA inhibitors;
* Known hypersensitivity to the study drug or excipients, known serious allergic reactions to any monoclonal antibody;
* Pulmonary artery invasion;
* History of leptomeningeal disease;
* Uncontrollable tumor-related pain;
* Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
* Uncontrolled or symptomatic hypercalcemia;
* Uncontrolled hypertension, history of hypertensive crisis or hypertensive encephalopathy;
* Patients with active autoimmune diseases, autoimmune diseases or systemic use of steroids/immunosuppressive agents;
* History of idiopathic pulmonary fibrosis, tissue pneumonia, drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on chest CT scan;
* Active pulmonary tuberculosis, or patients with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than 1 year ago but without regular treatment;
* Known human immunodeficiency virus (HIV) infection, active hepatitis B or C patients; HBsAg positive patients may participate in this study if HBV DNA testing is < 500 IU/ml or if the lower limit of detection at the site. HCV antibody positive patients may participate in this study if HCV RNA detection is less than the lower limit of detection value at the site where they are located;
* Patients with severe cardiovascular disease, such as New York Heart Association (NYHA) class 2 or higher heart failure, unstable angina pectoris, unstable arrhythmia, myocardial infarction or cerebrovascular accident within 6 months before enrollment;
* Patients with other malignant tumors (except for non-melanoma skin basal cell carcinoma or squamous cell carcinoma, breast/cervical carcinoma in situ, superficial bladder cancer and other carcinoma in situ who have received radical treatment and have no evidence of disease recurrence) within 5 years before the start of treatment or at the same time;
* According to the investigator 's judgment, the subject has other factors that may cause the subject to be forced to terminate the study halfway, such as having other serious diseases (including mental illness) requiring concomitant treatment, severely abnormal laboratory test values, and/or family or social factors that may affect the patient' s safety or collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicitys (DLTs) | up to 21 days after the first dose

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  Defined as the proportion of subjects achieving a complete response (CR) or partial response (PR) during treatment.
Disease control rate (DCR) | up to 2 years
  Defined as the proportion of subjects achieving complete response (CR) or partial response (PR) or stable disease (SD) during treatment.
Duration of response (DOR) | up to 2 years
  Defined as the time from the first documented response (CR or PR) to the first documented disease progression or death, whichever came first.
Progression-free survival (PFS) | up to 2 years
  Defined as the time from enrollment to the first documented disease progression or death from any cause, whichever came first.
Overall Survival (OS) | up to 2 years
  Defined as the time from enrollment to death due to any cause.

IPD SHARING:
Plan to Share IPD: No